CLINICAL TRIAL: NCT02593188
Title: Non-Interventional Post-Marketing Safety Study on the Long-Term Safety of HYQVIA (Global)
Status: Completed | Type: Observational
Sponsor: Baxalta now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Other Study IDs: 161406; EUPAS21523 (Registry Identifier: EU PAS)
Record Dates: First submitted 2015-10-29; First posted 2015-11-02 (Estimated); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Primary Immunodeficiency Diseases (PID)
MeSH Terms: conditions — Primary Immunodeficiency Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples (plasma) for antibodies against recombinant human hyaluronidase (rHuPH20) that remain after study testing will be stored at the Central Laboratory to confirm implausible or critical test results, if required. Samples will be stored in a coded form and according to local requirements for a maximum of 2 years after the final study report has been completed and subsequently will be destroyed.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HYQVIA- Epoch 1: Participants receiving HYQVIA
  Interventions: Biological: HYQVIA
- HYQVIA- Epoch 2: Participants with rHuPH antibody titers ≥160 (tested in Epoch 1)
  Interventions: Biological: HYQVIA

INTERVENTIONS:
Biological: HYQVIA — Immune Globulin Infusion 10% (Human) with Recombinant Human Hyaluronidase

SUMMARY:
The purpose of the proposed study is to acquire additional data (including the assessment of anti-rHuPH20 antibodies) on the long-term safety of HYQVIA and to assess the prescribed treatment regimens and treatment administration in routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Participant requires immunoglobulin treatment for primary immunodeficiency disease (PIDD)
2. Participant age is compatible with local package insert requirements
3. Participant has been prescribed or has started treatment with HYQVIA (Immune Globulin (Human) 10% with rHuPH20)
4. Participant is willing and able to comply with the requirements of the protocol.
5. Female participant of child-bearing potential agrees to inform the investigator if she becomes pregnant, or plans to become pregnant during the course of the study

Exclusion Criteria:

1. Participant has known hypersensitivity to any of the components of the medicinal product
2. Participant has participated in an interventional clinical study involving a medicinal product or device within 30 days prior to enrollment or is scheduled to participate in an interventional clinical study involving a medical product or device during the course of this study
3. Participant is a family member or employee of the investigator
4. Participant is planning to become pregnant, pregnant or breastfeeding at the time of enrollment

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2015-11-12 (Actual); Primary Completion 2021-10-21 (Actual); Study Completion 2021-10-21 (Actual)

PRIMARY OUTCOMES:
Incidence of all related serious adverse events (SAEs) | Throughout the study period of approximately 5 1/2 years
Incidence of all SAEs | Throughout the study period of approximately 5 1/2 years
Incidence of non-serious adverse events (AEs), related and not related, local and systemic. | Throughout the study period of approximately 5 1/2 years
Incidence of Infections | Throughout the study period of approximately 5 1/2 years
Incidence and titer of binding and neutralizing antibodies to rHuPH20 | Throughout the study period of approximately 5 1/2 years
Treatment Regimen: Total dose administered | Throughout the study period of approximately 5 1/2 years
Treatment Regimen: Infusion interval | Throughout the study period of approximately 5 1/2 years
Treatment Administration: Actual volume per infusion | Throughout the study period of approximately 5 1/2 years
Treatment Administration: Maximum infusion rate | Throughout the study period of approximately 5 1/2 years
Treatment Administration: Mean rate of infusion | Throughout the study period of approximately 5 1/2 years
Treatment Administration: Duration of infusion | Throughout the study period of approximately 5 1/2 years
Treatment Administration: Number of infusion sites per infusion | Throughout the study period of approximately 5 1/2 years
Health Related Quality of Life: Short Form-36 (SF-36) | Every 3 months in first year of study, annually for remainder of study
Health Related Quality of Life: EuroQol 5-Dimension (EQ-5D) Questionnaire | Every 3 months in first year of study, annually for remainder of study
Health Related Quality of Life: Treatment Satisfaction Questionnaire for Medication-9 (TSQM-9) | Every 3 months in first year of study, annually for remainder of study
Health Related Quality of Life: Treatment Preference Questionnaire | Annually throughout the study
Health resource use: hospitalizations | Throughout the study period of approximately 5 1/2 years
Health resource use: length of hospital stay | Throughout the study period of approximately 5 1/2 years
Health resource use: acute care visits | Throughout the study period of approximately 5 1/2 years
Health resource use: Emergency Room visits | Throughout the study period of approximately 5 1/2 years
Days missed from work/school | Throughout the study period of approximately 5 1/2 years

CONTACTS AND LOCATIONS:
Overall Officials: Shire Director, Study Director — Shire
Locations (30):
- United States (30):
  - Kern Allergy Medical Clinic, Bakersfield, California
  - University of California Irvine Medical Center, Irvine, California
  - Riviera Allergy Medical Center, Redondo Beach, California
  - Capital Allergy & Respiratory Disease Center, Sacramento, California
  - UCLA School of Medicine, Santa Monica, California
  - Asthma and Allergy Associates, PC, Colorado Springs, Colorado
  - Pikes Peak Allergy and Asthma, Colorado Springs, Colorado
  - IMMUNOe International Research Centers, Thornton, Colorado
  - Georgia Pollens Clinical Research Centers, Inc., Albany, Georgia
  - Boston Childrens Hospital, Boston, Massachusetts
  - Canton Health Center, Canton, Michigan
  - Washington University, St Louis, Missouri
  - Corning Center for Clinical Research, Corning, New York
  - Northwell Health, Inc. PRIME, Great Neck, New York
  - Winthrop University, Mineola, New York
  - Columbia University Medical Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Carolinas Healthcare System, Charlotte, North Carolina
  - Allergy Asthma & Immunology Relief of Charlotte, Charlotte, North Carolina
  - Optimed Research, LTD, Columbus, Ohio
  - Allergy, Asthma and Clinical Research Center, Oklahoma City, Oklahoma
  - OK Institute of Allergy & Asthma Clinical Research, LLC, Oklahoma City, Oklahoma
  - Vital Prospects Clinical Research Institute, P.C., Tulsa, Oklahoma
  - Allergy & Clinical Immunology Associates, Pittsburgh, Pennsylvania
  - National Allergy, Asthma & Urticaria Centers of Charleston, PA, North Charleston, South Carolina
  - Allergy / Immunology Research Center of North Texas, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas
  - McKinney Allergy and Asthma Center, McKinney, Texas
  - Greater Austin Allergy, Asthma, & Immunology, Round Rock, Texas
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link. — https://clinicaltrials.takeda.com/study-detail/5f6b5fc54db2bf003ab45c45?idFilter=%5B%22161406%22%5D